CLINICAL TRIAL: NCT02056561
Title: Investigation Of The Effects Of General Anesthesia On The Oxidant/Antioxidant System
Brief Title: Effects on Immun System of Anesthesia
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, yavuz demiraran, Professor Doctor, Duzce University
Other Study IDs: MESUT-81
Record Dates: First submitted 2014-01-29; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Anesthesia
Keywords: Anesthesia; Oxidants; Antioxidants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — Before induction and after the operation venous blood samples were taken.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- TIVA (group T n: 15): Group T were given propofol infusions of 12 mg/kg/hr for the first 10 minutes, 9 mg/kg/hr for the second 10 minutes and 6 mg/kg/hr after that. Patients were ventilated with 50% air and 50% O2 mix at 6 L/min flow.
- Sevoflurane (group S n: 15): Group S were ventilated with 2% sevoflurane, 50% air and 50% O2 mix at 6 L/min flow.
- Desflurane (group D n: 15): Group D cases were given 6% desflurane 50% air and 50% O2 mix at 6 L/min flow.

SUMMARY:
Introduction and Aim: Desflurane and sevoflurane are frequently used for maintenance of anesthesia and studies have shown that these anesthetics cause a variety of changes in oxidative stress and antioxidative defense mechanisms. The chemical structure of propofol is similar to some free radical consumers such as endogenous vitamin E and butylated hydroxene toluene. This study aims to compare the effects of sevoflurane, desflurane and propofol infusion anesthesia on the oxidant and antioxidant systems of patients undergoing laparoscopic cholecystectomy.

Material and Method: Forty-five patients, ASA (American Society of Anesthesiologists) I-II, score between 18-50 years with planned laparoscopic cholecystectomy under general anesthesia were included in the study. Patients were divided into 3 groups as total intravenous anesthesia (TIVA) (group T n: 15), sevoflurane (group S n: 15) and desflurane (group D n: 15). Propofol 2 mg/kg IV, fentanyl 1 mcg/kg IV, vecuronium 0.1 mg/kg IV given to all groups for anesthesia induction. For maintenance of anesthesia group S were ventilated with 2% sevoflurane, 50% air and 50% O2 mix at 6 L/min flow. Group D were given 6% desflurane 50% air and 50% O2 mix at 6 L/min flow. Group T were given propofol infusions of 12 mg/kg/hr for the first 10 minutes, 9 mg/kg/hr for the second 10 minutes and 6 mg/kg/hr after that. Patients were ventilated with 50% air and 50% O2 mix at 6 L/min flow. Before induction and after the operation venous blood samples were taken to evaluate the levels of glutathion peroxidase, total oxidants and antioxidants.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II with patients
* Between 18-50 years
* Planned laparoscopic cholecystectomy under general anesthetic

Exclusion Criteria:

* Patients with endocrine dysfunction
* blood transfusion in the previous 2 weeks
* signs of infection and inflammation
* history of preoperative medication use
* anemia
* hemorrhage requiring transfusion during the operation were excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 45 patients ASA I-II between 18-50 years with planned laparoscopic cholecystectomy under general anesthetic were included in the study. Patients were divided into 3 groups on the way to surgery; TIVA (group T n: 15), sevoflurane (group S n: 15) and desflurane (group D n: 15).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Levels of glutathion peroxidase, total oxidants and antioxidants. | 24 hours
  Before induction and after the operation venous blood samples were taken to evaluate the levels of glutathion peroxidase, total oxidants and antioxidants.

CONTACTS AND LOCATIONS:
Overall Officials: yavuz demiraran, MD prof, Principal Investigator — duzce university medical faculty
Locations (1):
- Duzce Univercity Medical Fauculty, Düzce, Turkey (Türkiye)